CLINICAL TRIAL: NCT00956839
Title: Double-blind Randomized Study to Determine the Efficacy of Intramuscular Vitamin D3 Supplementation in Tropical Calcific Pancreatitis
Brief Title: Prospective Study of Efficacy of Intra-muscular Vitamin D3 in Tropical Calcific Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Eesh Bhatia, Doctor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/AA/EMP/IEC/46/25.7.09
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatitis, Chronic
Keywords: Tropical calcific pancreatitis; Tropical chronic pancreatitis; Chronic pancreatitis; Vitamin D; Vitamin D deficiency; Cholecalciferol; Intramuscular vitamin D3
MeSH Terms: conditions — Pancreatitis, Chronic; Tropical Calcific Pancreatitis; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): IM Vitamin D3 3,00,000 Units single dose
  Interventions: Drug: Vitamin D3 (Cholecalciferol)
- Group B (Active Comparator): IM vitamin D3 6,00,000 Units single dose
  Interventions: Drug: Vitamin D3 (Cholecalciferol)
- Group C (Active Comparator): Oral vitamin D3 500 Units/ day
  Interventions: Drug: Vitamin D3 (Cholecalciferol)

INTERVENTIONS:
Drug: Vitamin D3 (Cholecalciferol) — Arm 1 - Intramuscular vitamin D3 3,00,000 Units single dose
  Arm 2 - Intramuscular vitamin D3 6,00,000 Units single dose
  Arm 3 - Oral vitamin D3 500 Units/day for 6 months
  Other Names: IM vitamin D3 - Inj Arachitol (Solvay, India); Oral vitamin D3 - Tab Cipcal (Cipla, India)

SUMMARY:
The purpose of this study is to determine the efficacy of 2 different doses of intramuscular (IM) vitamin D3 as compared to an oral replacement dose in normalizing vitamin D levels in the blood of patients with tropical calcific pancreatitis.

DETAILED DESCRIPTION:
Tropical calcific pancreatitis (TCP) is a form of chronic pancreatitis unique to developing countries. Patients with TCP often have malabsorption leading to nutritional deficiencies. We have noted that vitamin D deficiency is common in patients with TCP. The ideal regimen for supplementing vitamin D3 in chronic pancreatitis remains unclear and there are no previous studies available. High dose oral vitamin D2 has been shown to be ineffective in normalizing vitamin D levels in patients with pancreatic insufficiency due to cystic fibrosis.

Intramuscular (IM) vitamin D3 supplementation in chronic pancreatitis has certain advantages. Firstly, decreased and inconsistent absorption from the intestine is avoided. Secondly, IM vitamin D3 has a long duration of action (6-12 months). The safety of high-dose IM vitamin D3 has been proven in previous studies in healthy individuals. Finally, the injection form is considerably less expensive as compared to oral vitamin D3.

The aim of the current prospective double blind study is to compare 2 regimens of high dose IM vitamin D3 replenishment with oral vitamin D3 in standard recommended doses in normalizing serum vitamin D3 levels in patients with TCP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of tropical calcific pancreatitis established by history of abdominal pain or diabetes and evidence on ultrasound or CT scan of pancreatic ductal dilatation and intra-ductal stones

Exclusion Criteria:

* History of alcohol intake or any secondary cause for chronic pancreatitis (hypercalcemia, hypertriglyceridemia, biliary tract stones)
* History of hepatic or renal dysfunction or of current intake of drugs such as steroids, anticonvulsant drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eesh Bhatia, MD, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, India
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Background] Mann ST, Stracke H, Lange U, Klor HU, Teichmann J. Vitamin D3 in patients with various grades of chronic pancreatitis, according to morphological and functional criteria of the pancreas. Dig Dis Sci. 2003 Mar;48(3):533-8. doi: 10.1023/a:1022540816990. PMID 12757166
- [Background] Barman KK, Premalatha G, Mohan V. Tropical chronic pancreatitis. Postgrad Med J. 2003 Nov;79(937):606-15. doi: 10.1136/pmj.79.937.606. PMID 14654569
- [Background] Dujsikova H, Dite P, Tomandl J, Sevcikova A, Precechtelova M. Occurrence of metabolic osteopathy in patients with chronic pancreatitis. Pancreatology. 2008;8(6):583-6. doi: 10.1159/000159845. Epub 2008 Sep 29. PMID 18824882
- [Background] Aris RM, Merkel PA, Bachrach LK, Borowitz DS, Boyle MP, Elkin SL, Guise TA, Hardin DS, Haworth CS, Holick MF, Joseph PM, O'Brien K, Tullis E, Watts NB, White TB. Guide to bone health and disease in cystic fibrosis. J Clin Endocrinol Metab. 2005 Mar;90(3):1888-96. doi: 10.1210/jc.2004-1629. Epub 2004 Dec 21. PMID 15613415
- [Background] Boyle MP, Noschese ML, Watts SL, Davis ME, Stenner SE, Lechtzin N. Failure of high-dose ergocalciferol to correct vitamin D deficiency in adults with cystic fibrosis. Am J Respir Crit Care Med. 2005 Jul 15;172(2):212-7. doi: 10.1164/rccm.200403-387OC. Epub 2005 Apr 28. PMID 15860755
- [Background] Green D, Carson K, Leonard A, Davis JE, Rosenstein B, Zeitlin P, Mogayzel P Jr. Current treatment recommendations for correcting vitamin D deficiency in pediatric patients with cystic fibrosis are inadequate. J Pediatr. 2008 Oct;153(4):554-9. doi: 10.1016/j.jpeds.2008.04.058. Epub 2008 Jun 27. PMID 18589445
- [Background] Lark RK, Lester GE, Ontjes DA, Blackwood AD, Hollis BW, Hensler MM, Aris RM. Diminished and erratic absorption of ergocalciferol in adult cystic fibrosis patients. Am J Clin Nutr. 2001 Mar;73(3):602-6. doi: 10.1093/ajcn/73.3.602. PMID 11237938
- [Background] Diamond TH, Ho KW, Rohl PG, Meerkin M. Annual intramuscular injection of a megadose of cholecalciferol for treatment of vitamin D deficiency: efficacy and safety data. Med J Aust. 2005 Jul 4;183(1):10-2. doi: 10.5694/j.1326-5377.2005.tb06879.x. PMID 15992330
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Derived] Reddy SV, Ramesh V, Bhatia E. Double blind randomized control study of intramuscular vitamin D3 supplementation in tropical calcific pancreatitis. Calcif Tissue Int. 2013 Jul;93(1):48-54. doi: 10.1007/s00223-013-9726-6. Epub 2013 Apr 6. PMID 23564348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Endocrinology and Gastroenterology Clinics of Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow from July 2009 to December 2009
Pre-assignment Details: All patients who consented for the study were enrolled and randomized.
Groups:
- IM Vitamin D3 3,00,000 Units: IM Vitamin D3 3,00,000 Units single dose
- IM Vitamin D3 6,00,000 Units: IM vitamin D3 6,00,000 Units single dose
- Oral Vitamin D3: Oral vitamin D3 500 Units/ day
Period: Overall Study
Arm/Group | IM Vitamin D3 3,00,000 Units | IM Vitamin D3 6,00,000 Units | Oral Vitamin D3
Started | 14 | 13 | 13
Completed | 11 | 13 | 10
Not Completed | 3 | 0 | 3
Not completed — Lost to Follow-up | 3 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Vitamin D3 3,00,000 Units | IM Vitamin D3 6,00,000 Units | Oral Vitamin D3 | Total
Number analyzed (Participants) | 14 | 13 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 40
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.9) | 33.9 (10.6) | 34.3 (9.2) | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 14
  Male | 8 | 10 | 8 | 26
Region of Enrollment [Number; unit: participants]
  India | 14 | 13 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Serum 25 Hydroxy Vitamin D3 > 30 ng/ml
Description: Percentage of patients in each group with serum 25 hydroxy vitamin D >30 ng/ml
Time Frame: 6 months post intervention
Population: Intention to treat analysis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | IM Vitamin D3 3,00,000 Units | IM Vitamin D3 6,00,000 Units | Oral Vitamin D3
Number analyzed (Participants) | 14 | 13 | 13
percentage of patients | 85 [75.1 to 94.9] | 29 [16.9 to 41.1] | 0 [0 to 0]

2. Secondary Outcome: Serum Total Calcium
Description: Serum total calcium (mg/dL) at time points 0, 1, 3 and 6 months
Time Frame: 0, 1, 3, 6 months post intervention
Population: at time points 0, 1, 3 and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IM Vitamin D3 3,00,000 Units | IM Vitamin D3 6,00,000 Units | Oral Vitamin D3
Number analyzed (Participants) | 14 | 13 | 13
mg/dL
  baseline | 9.20 (0.48) [0 to 0] | 9.56 (0.48) [0 to 0] | 9.24 (0.48) [0 to 0]
  1 month | 9.28 (0.44) | 9.52 (0.40) | 9.28 (0.52)
  3 months | 9.40 (0.52) | 9.44 (0.48) | 9.40 (0.52)
  6 months | 9.40 (0.60) | 9.40 (0.60) | 9.28 (0.48)

ADVERSE EVENTS:
Arm/Group | IM Vitamin D3 3,00,000 Units | IM Vitamin D3 6,00,000 Units | Oral Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes